CLINICAL TRIAL: NCT01315002
Title: Nicotine Effects on Endophenotypes of Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: Principal Investigator, Nadine Petrovsky, PhD, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NICSZ001; 2008-001362-90 (EudraCT Number)
Record Dates: First submitted 2011-03-14; First posted 2011-03-15 (Estimated); Results first posted 2015-01-16 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Schizophrenia
Keywords: nicotine; schizophrenia; endophenotype
MeSH Terms: conditions — Schizophrenia | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotine Patch (Active Comparator): Transdermal nicotine patch
  Interventions: Drug: Transdermal nicotine patch
- Placebo patch (Placebo Comparator): Placebo patch
  Interventions: Drug: Placebo patch

INTERVENTIONS:
Drug: Transdermal nicotine patch — 7mg transdermal nicotine patch (non-smoking subjects) 14mg transdermal nicotine patch (smoking subjects)
  Other Names: NiQuitin Clear, GlaxoSmithKline Germany
  Arms: Nicotine Patch
Drug: Placebo patch — Placebo patch
  Other Names: band-aid by Fink and Walter GmbH, Germany
  Arms: Placebo patch

SUMMARY:
The purpose of this study is to test the effects of nicotine on cognition with the following schizophrenia endophenotypes: prepulse inhibition, antisaccades, the continuous performance test, spatial working memory and a verbal memory task. Schizophrenia patients, unaffected first-degree relatives of schizophrenia patients and healthy controls receive transdermal nicotine in a double-blind, placebo-controlled, crossover study.

DETAILED DESCRIPTION:
Convergent findings suggest that an altered neuronal nicotinic acetylcholine receptor system may contribute to the pathophysiology of schizophrenia. Nicotine consumption through cigarette smoking might represent a form of self-medication in schizophrenia as nicotine reduces cognitive and physiological deficits in schizophrenia. The present study aims to investigate how nicotine affects attentional and executive schizophrenia endophenotypes and how genetic polymorphisms relating to the cholinergic system might play a role in inter-individual differences in the magnitude of nicotine effects.

Schizophrenia patients, first-degree relatives of schizophrenia patients as well as healthy controls will receive transdermal nicotine in a double-blind, placebo-controlled, crossover study and will be assessed with prepulse inhibition, antisaccades, the continuous performance test, spatial working memory and a verbal memory task. Subjects will be overnight-abstinent smokers and non-smokers. However, the investigators will particularly test non-smokers in order to eliminate confounding effects of nicotine withdrawal and reinstatement.

Main hypotheses:

* Schizophrenia patients will perform worse than matched controls in all cognitive tests (validating our endophenotypes).
* Nicotine administration will enhance cognitive performance in overnight-abstinent smokers.
* Improvement of cognitive performance in smokers with schizophrenia will be stronger than in control smokers.
* Improvement of cognitive performance in smoking first-degree relatives of schizophrenia patients will be stronger than in control smokers.
* Nicotine administration will affect cognitive functioning in non-smoking subjects.
* Nicotine administration will improve cognitive functioning in non-smoking schizophrenia patients.
* The effects of nicotine in non-smoking subjects are stronger in those subjects who are cognitively more impaired (i.e. performing below the median of the respective group).

The present research contributes to the issue whether nicotinic cholinergic receptor agonists may have therapeutic value in the treatment of cognition in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM IV) diagnosis of schizophrenia
* age 18-55 years old
* able to provide informed consent
* treated with antipsychotic medications at a stable dose for at least 6 weeks
* normal or corrected to normal vision
* smokers (Fagerström Test for Nicotine Dependence > 4)
* non-smokers (< 100 cigarettes/lifetime, not having smoked in the past year)

Controls:

* age 18-55 years old
* able to provide informed consent
* normal or corrected to normal vision
* smokers (Fagerström Test for Nicotine Dependence > 4)
* non-smokers (< 100 cigarettes/lifetime, not having smoked in the past year)

Unaffected First-Degree Relatives of Schizophrenia Patients:

* same inclusion criteria as controls plus
* having an adult first-degree relative (sibling, parent, child) with a DSM IV diagnosis of schizophrenia

Exclusion Criteria:

Patients:

* substance dependence
* clinical instability
* changes in medication in the last 6 weeks
* anticholinergic medication
* untreated hypertension
* cardiovascular disease
* insulin-dependent diabetes mellitus
* phaeochromocytoma
* uncontrolled hyperthyroidism
* renal or hepatic impairment
* central nervous system disease
* pulmonary disease
* generalised dermatological disorders (neurodermatitis, psoriasis, chronic dermatitis, urticaria, etc.)
* gastric or intestinal ulcer
* hypersensitivity to nicotine
* allergy to patches
* women: pregnancy, lactation

Controls:

* substance dependence
* having a first-, second-, or third-degree relative with a psychotic disorder
* DSM IV Axis I disorder
* anticholinergic medication
* untreated hypertension
* cardiovascular disease
* insulin-dependent diabetes mellitus
* phaeochromocytoma
* uncontrolled hyperthyroidism
* renal or hepatic impairment
* central nervous system disease
* pulmonary disease
* generalised dermatological disorders (neurodermatitis, psoriasis, chronic dermatitis, urticaria, etc.)
* gastric or intestinal ulcer
* hypersensitivity to nicotine
* allergy to patches
* women: pregnancy, lactation

Unaffected First-Degree Relatives of Schizophrenia Patients:

* same exclusion criteria as controls

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2008-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wagner, Prof. Dr., Principal Investigator — University Hospital, Bonn; Wolfgang Maier, Prof. Dr., Principal Investigator — University Hospital, Bonn

RESULTS

PARTICIPANT FLOW:
Groups:
- Nicotine First, Then Placebo: Transdermal nicotine patch first (single application), then placebo patch (single application, one week after administration of nicotine patch)
  Doses:
  non-smokers: 7mg transdermal nicotine patch smokers: 14mg transdermal nicotine patch
- Placebo First, Then Nicotine: Placebo patch first (single application), then transdermal nicotine patch (single application, one week after administration of placebo patch)
  Doses:
  non-smokers: 7mg transdermal nicotine patch smokers: 14mg transdermal nicotine patch
Period: Overall Study
Arm/Group | Nicotine First, Then Placebo | Placebo First, Then Nicotine
Started | 61 | 60
Completed | 56 | 55
Not Completed | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Includes groups randomized to receive nicotine first and placebo first. Number of all study participants = 121.
Arm/Group | All Study Participants
Number analyzed (Participants) | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 121
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.23 (9.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 68
Region of Enrollment [Number; unit: participants]
  Germany | 121

OUTCOME MEASURES:

1. Primary Outcome: Error Percentage in Antisaccade Task
Description: Three hours after the application of a nicotine or a placebo patch, performance on the antisaccade task is assessed. In the antisaccade task participants visually fixate a central stimulus which is replaced by a sudden onset target that appears at some distance to the left or right. Participants are told to refrain from looking at the peripheral target, and direct their gaze instead in the opposite direction (i.e. they have to make an antisaccade). Participants typically fail to achieve this on a significant number of trials and instead make reflexive glances towards the target (i.e. making a so-called antisaccade error). Error percentage in the antisaccade task is the unit of measure in this task. Error percentage in the antisaccade task = number of antisaccade errors / total number of trials.
Time Frame: Three hours after patch application
Measure: Mean (Standard Deviation); unit: Error Percentage in Antisaccade Task
Arm/Group | Nicotine Patch | Placebo Patch
Number analyzed (Participants) | 111 | 111
Error Percentage in Antisaccade Task | 22.6 (17.0) | 29.1 (19.1)
Statistical Analysis 1: Comparison: Nicotine Patch vs Placebo Patch; Null hypothesis is that there was no difference in change of error percentage in the antisaccade task between nicotine and placebo. An ANOVA model was used with treatment (nicotine, placebo) as a within-subjects factor. The test was performed with a significance level of 0.05 (two-sided). Results showed significantly better antisaccade performance (i.e. less antisaccade errors) in the nicotine condition; Test type: Superiority or Other; p < 0.05, ANOVA

ADVERSE EVENTS:
Time Frame: 3 years, 8 months
Arm/Group | Nicotine First, Then Placebo | Placebo First, Then Nicotine
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/60
Other Adverse Events (participants affected / at risk) | 5/61 | 5/60
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nicotine First, Then Placebo (N=61) | Placebo First, Then Nicotine (N=60)
Nausea (Gastrointestinal disorders) | 2 | 4
Vomiting (Gastrointestinal disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes